CLINICAL TRIAL: NCT07190508
Title: The Effects of Pre-Sedation Fluid Replacement and Endoscopic Duodenal Passage on Intraocular Pressure: A Prospective Observational Study
Brief Title: Pre-Sedation Fluid Replacement and Duodenal Passage Effects on Intraocular Pressure
Acronym: ENDO-IOP
Status: Completed | Type: Observational
Sponsor: Sevim Şenol Karataş (Other)
Responsible Party: Sponsor-Investigator, Sevim Şenol Karataş, Specialist in Anesthesiology, Elazıg Fethi Sekin Sehir Hastanesi
Organization: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Other Study IDs: EFSH-ANES-2025-09-IOP
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Intraocular Pressure Changes; Upper Gastrointestinal Endoscopy
Keywords: Intraocular Pressure; Endoscopy, Gastrointestinal; Sedation; Propofol; Midazolam; Fentanyl; Duodenum; Tonometer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Upper GI Endoscopy Patients: Adult patients (≥18 years) undergoing diagnostic upper gastrointestinal endoscopy with standard pre-sedation isotonic fluid replacement and sedoanalgesia. Intraocular pressure is measured at four predefined time points: baseline, after fluid replacement, after sedoanalgesia, and after duodenal intubation.
  Interventions: Other: No Intervention (Observational)

INTERVENTIONS:
Other: No Intervention (Observational) — Participants undergo routine diagnostic upper gastrointestinal endoscopy with standard institutional care. No additional intervention is applied beyond usual clinical practice.

SUMMARY:
This prospective observational study investigates whether routine pre-sedation isotonic fluid replacement and the passage of the endoscope into the duodenum acutely affect intraocular pressure (IOP) in adult patients undergoing diagnostic upper gastrointestinal endoscopy. A non-contact tonometer is used to measure IOP at four predefined time points: baseline, after pre-sedation fluid replacement, after sedoanalgesia, and immediately following duodenal intubation. Hemodynamic parameters, oxygen saturation, and sedative doses are also recorded. The primary aim is to determine changes in IOP during the procedure, while secondary outcomes include the relationship between hemodynamic fluctuations, sedative requirements, and IOP changes. The findings are expected to provide insights into the safety of endoscopy with respect to ocular physiology, particularly in patients at risk of increased intraocular pressure.

DETAILED DESCRIPTION:
This single-center, prospective, observational cohort study is conducted at Elazig Fethi Sekin City Hospital, Türkiye. The study population consists of adults (≥18 years) scheduled for diagnostic upper gastrointestinal endoscopy under routine sedoanalgesia. Consecutive eligible patients are enrolled until the target sample size of 40 is reached. Exclusion criteria include any history of glaucoma, ocular surgery, or ongoing ophthalmological treatment.

All participants receive standard pre-sedation isotonic fluid replacement (500 mL) as per institutional protocol. Sedoanalgesia is administered with propofol, midazolam, and fentanyl at the discretion of the attending anesthesiologist, following routine practice. Intraocular pressure (IOP) is measured using a calibrated non-contact tonometer at four time points: (1) baseline before fluid loading, (2) after fluid replacement and before sedation, (3) after sedoanalgesia, and (4) immediately following duodenal intubation. Measurements are consistently taken from the same eye and patient position to ensure reliability.

In addition to IOP, systolic/diastolic blood pressure, mean arterial pressure, heart rate, and peripheral oxygen saturation are continuously monitored and recorded. Sedative drug doses and procedure times (total duration and time to duodenal passage) are documented. The primary outcome is the change in IOP between baseline and post-duodenal intubation. Secondary outcomes include correlations between hemodynamic variables, sedative consumption, and intraocular pressure changes, as well as subgroup analyses according to age, sex, and comorbidities.

Statistical analysis will include repeated-measures ANOVA or non-parametric equivalents to compare IOP at different time points, along with regression models to identify predictors of IOP changes. With a sample size of at least 34 patients (allowing for 40 to compensate for dropouts), the study has adequate power to detect clinically significant differences.

The results are expected to contribute to a better understanding of the physiological ocular effects of upper GI endoscopy and to inform clinical practice, especially in patients at risk of elevated intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Scheduled for diagnostic upper gastrointestinal endoscopy under sedoanalgesia
* ASA physical status I-III
* Voluntarily provides informed consent

Exclusion Criteria:

* History of glaucoma or ocular hypertension
* Previous ocular surgery or ongoing ophthalmological treatment
* Known contraindications to sedoanalgesia (propofol, midazolam, fentanyl)
* ASA physical status IV or higher

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) scheduled for diagnostic upper gastrointestinal endoscopy under sedoanalgesia at Elazig Fethi Sekin City Hospital. Consecutive eligible patients will be approached and enrolled after providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) | During the procedure (baseline, after fluid replacement, after sedoanalgesia, and immediately after duodenal intubation; total duration ≈ 30 minutes)
  IOP is measured using a calibrated non-contact tonometer at four predefined time points: baseline, after isotonic fluid replacement, after sedoanalgesia, and after endoscopic duodenal passage. Measurements are obtained from the same eye in the same patient position to ensure consistency.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) | During the procedure (baseline, after fluid replacement, after sedoanalgesia, and after duodenal intubation; ~30 minutes)
  Systolic blood pressure will be recorded continuously at each predefined time point.
Change in Diastolic Blood Pressure (DBP) | During the procedure (baseline, after fluid replacement, after sedoanalgesia, and after duodenal intubation; ~30 minutes)
  Diastolic blood pressure will be recorded continuously at each predefined time point.
Change in Mean Arterial Pressure (MAP) | During the procedure (baseline, after fluid replacement, after sedoanalgesia, and after duodenal intubation; ~30 minutes)
  Mean arterial pressure will be recorded continuously at each predefined time point.
Change in Heart Rate (HR) | During the procedure (baseline, after fluid replacement, after sedoanalgesia, and after duodenal intubation; ~30 minutes)
  Heart rate will be recorded continuously at each predefined time point.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Şenol Karataş, MD, Principal Investigator — Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study is a single-center observational project with a limited sample size and no data repository plan. Only aggregated results will be reported in publications.

REFERENCES:
- [Background] Berdahl JP, Allingham RR, Johnson DH. Cerebrospinal fluid pressure is decreased in primary open-angle glaucoma. Ophthalmology. 2008 May;115(5):763-8. doi: 10.1016/j.ophtha.2008.01.013. PMID 18452762
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- See also: Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation — https://elazigsehir.saglik.gov.tr/